CLINICAL TRIAL: NCT02203565
Title: Pilot Study to Investigate the Impact of Hypochlorite in the Prevention of Radiation Dermatitis
Brief Title: Dakin's Solution in Preventing Radiation Dermatitis in Patients With Breast Cancer Undergoing Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kathleen Horst, Assistant Professor of Radiation Oncology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BRS0039; NCI-2014-01551 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB-29833; BRS0039 (Other: OnCore); P30CA124435 (NIH)
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer; Skin Reactions Secondary to Radiation Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Sodium Hypochlorite; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive care (Dakin's solution, radiation therapy) (Experimental): Patients apply Dakin's solution topically daily over 10 minutes within 60 minutes of radiation therapy for up to 6 weeks.
  Interventions: Drug: Dakin's solution; Radiation: radiation therapy; Other: questionnaire administration; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: Dakin's solution — Applied topically
  Other Names: aqueous solution of sodium hypochlorite; Dakin's fluid
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Other: questionnaire administration — Ancillary studies
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
This pilot clinical trial studies Dakin's solution in preventing radiation dermatitis in patients with breast cancer undergoing radiation therapy. Radiation dermatitis is a skin condition in which the affected skin becomes painful, red, itchy, and blistered. Dakin's solution may help reduce dermatitis caused by radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the percent change in women who experience grade 3 or 4 radiation dermatitis as defined by the Stanford Radiation Dermatitis Scoring System during radiation treatment for breast cancer compared to historical experience using standard skin care.

SECONDARY OBJECTIVES:

I. To assess the feasibility of daily application of the hypochlorite solution (Dakin's solution), and to assess levels of pain during radiotherapy treatment.

OUTLINE:

Patients apply Dakin's solution topically daily over 10 minutes within 60 minutes of radiation therapy for up to 6 weeks.

After completion of study treatment, patients are followed up at 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women with breast cancer who plan to undergo radiation therapy to the breast or chest wall
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Women with scleroderma or discoid lupus
* Women with inflammatory breast cancer as evidenced by clinical assessment
* Women with breast cancer involving the skin
* Women who have undergone prior radiotherapy to the chest wall and/or breast

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07-07 (Actual); Study Completion 2016-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Horst, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supportive Care (Dakin's Solution, Radiation Therapy)
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care (Dakin's Solution, Radiation Therapy)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Percent of Women Who Develop Grade 3 or 4 Radiation Dermatitis (as Defined by the Stanford Radiation Dermatitis Scoring System) During a Course of Radiation Therapy
Description: Stanford Radiation Dermatitis Scoring System:
  Grade Clinical finding
  0 No skin change
  1 Faint, barely detectable erythema 2 Follicular rash, hyperpigmentation, evolving erythema 3 Dry desquamation, brisk erythema 4 Moist desquamation 5 Bleeding, ulceration, and/or infection
Time Frame: Baseline to up to 6 weeks after completion of therapy
Population: Patients with complete data for analysis. While 20 patients were enrolled in the study, only 14 had data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Dakin's Solution, Radiation Therapy)
Number analyzed (Participants) | 14
Participants | 6

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout radiation treatment, approximately 5 weeks, for each patients. For the study overall adverse events were monitored for various patients over the course of 1 year when the study was open to accrual.
Arm/Group | Supportive Care (Dakin's Solution, Radiation Therapy)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Dakin's Solution, Radiation Therapy) (N=20)
Dermatitis radiation (Skin and subcutaneous tissue disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Dakin's Solution, Radiation Therapy) (N=20)
Radiation Dermatitis (Skin and subcutaneous tissue disorders) | 20 (20) — Patients were evaluated for Radiation Dermatitis of all grades (1-4) as defined by CTCAE guidlines. Radiation dermatitis is an expected side effect of radiation therapy and not associated with or an expected reaction to the Dakin's solution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No